CLINICAL TRIAL: NCT04227275
Title: A Phase 1 Open-Label, Multi-Center Study of PSMA Targeted Genetically Modified Chimeric Antigen Receptor T Cells in Patients With Metastatic Castration Resistant Prostate Cancer
Brief Title: A Study of CART-PSMA-TGFβRDN in Patients With Metastatic Castration Resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Based on the safety events and evidence of biologic activity without sustained clinical responses the Sponsor finds the risk/benefit analysis unfavorable for patients and has terminated the study.
Sponsor: Tceleron Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CART-PSMA-TGFβRDN-02
Record Dates: First submitted 2019-12-12; First posted 2020-01-13 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Chimeric Antigen Receptor (CAR); T-cells; Prostate-Specific Membrane Antigen (PSMA); Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cyclophosphamide; fludarabine; Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Intervention Model Description: Sequential dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): Dose escalation of intravenous CART-PSMA-TGFβRDN cells for patients with metastatic castration resistant prostate cancer
  Interventions: Biological: CART-PSMA-TGFβRDN; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Anakinra

INTERVENTIONS:
Biological: CART-PSMA-TGFβRDN — Intravenous administration of genetically modified autologous T cells engineered to express a protein capable of recognizing the tumor antigen prostate-specific membrane antigen (PSMA), as well as a dominant negative TGFβ receptor
Drug: Cyclophosphamide — Patients will receive cyclophosphamide and fludarabine lymphodepletion chemotherapy followed by the investigational product, CART-PSMA-TGFβRDN genetically modified T cells
Drug: Fludarabine — Patients will receive cyclophosphamide and fludarabine lymphodepletion chemotherapy followed by the investigational product, CART-PSMA-TGFβRDN genetically modified T cells
Drug: Anakinra — In applicable cohorts, patients will receive anakinra prophylactically starting on the day of administration of investigational product, CART-PSMA-TGFβRDN genetically modified T cells

SUMMARY:
Multi-center, open-label, Phase 1 study of the safety, tolerability and feasibility of dosing patients harboring metastatic castration resistant prostate cancer (mCRPC) with genetically modified autologous T cells (CART-PSMA-TGFβRDN cells) engineered to express a chimeric antigen receptor (CAR) capable of recognizing the tumor antigen prostate-specific membrane antigen (PSMA) and activating the T cell.

DETAILED DESCRIPTION:
This is a Phase 1 single-arm study designed to identify the dose and regimen of CART-PSMA- TGFβRDN cells that can be safely administered intravenously following the lymphodepletion (LD) regimen to patients with metastatic castration resistant prostate cancer (mCRPC). Following Dose Escalation, a Cohort Expansion will enroll patients to further explore the safety and tolerability of the selected dose and schedule.

It is anticipated that up to 50 patients will enroll in this study in both dose escalation and cohort expansion.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed histologic diagnosis of prostate cancer and have mCRPC, with castrate levels of testosterone (<50 ng/mL)
* PSA measurable disease per Prostate Working Group 3 (PCWG3) criteria
* Prior therapies defined as at least 2 prior lines of systemic therapy for prostate cancer, including at least one second generation androgen receptor inhibitor and/or CYP17α inhibitor. At least one line of prior therapy must be in the mCRPC setting
* Estimated estimated glomerular filtration rate ≥ 60 mL/min by Modification of Diet in Renal Disease criteria
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5x the upper limit of normal (ULN); patients with hepatic metastases ALT and AST ≤ 3.0 x ULN
* Serum total bilirubin < 1.5 mg/dL unless patient has known Gilbert's Syndrome, then serum bilirubin ≤3 mg/dL
* Serum albumin ≥ 3.0 g/dL
* Left ventricular ejection fraction (LVEF) ≥ 50%. LVEF assessment must have been performed within 8 weeks of enrollment
* Hemoglobin ≥ 8 g/dL
* Absolute neutrophil count ≥ 1000/μL
* Platelet count ≥ 75,000/μL
* Patients who have not undergone bilateral orchiectomy must be able to continue gonadotropin-releasing hormone (GnRH) therapy during the study
* Eastern Cooperative Oncology Group (ECOG) score of 0 or 1
* Toxicities from any previous therapy must have recovered to Grade 1 or baseline
* Patients of reproductive potential agree to use of approved highly effective contraceptive methods

Exclusion Criteria:

* Active invasive cancer, other than the proposed cancer included in the study, within 2 years prior to screening, unless treated with curative intent
* Current treatment with systemic corticosteroids (defined as a dose greater than the equivalent of prednisone 10 mg/day)
* Active autoimmune disease (including connective tissue disease, uveitis, sarcoidosis, inflammatory bowel disease or multiple sclerosis) or a history of severe autoimmune disease requiring prolonged immunosuppressive therapy (any immunosuppressive therapy within 6 weeks prior to screening visit)
* Current human immunodeficiency virus (HIV), hepatitis C virus, hepatitis B virus infections; Patients who are hepatitis B core antigen positive, hepatitis B surface antigen negative, should have a quantitative viral load measured; If viral load is undetectable, the patient will not be excluded if hey are able to be treated with anti-viral medication for at least 7 days prior to lymphodepletion until at least 6 months after infusion with viral load and ALT monitoring
* Active or uncontrolled medical or psychological condition that would preclude participation
* History of seizure disorder
* Prior allogeneic stem cell transplant
* Central nervous system malignancy
* History of severe infusion reaction to monoclonal antibodies or biological therapies, or to study product excipients that would preclude the patient safely receiving CART-PSMA-TGFβRDN cells
* History of being previously treated with a J591 antibody-based therapy
* Ferritin levels ≥ 4x the upper limit of normal prior to apheresis or prior to the start of lymphodepleting chemotherapy
* Active or recent (within the past 6 months prior to apheresis or lymphodepletion) cardiovascular disease, defined as (1) New York Heart Association Class III or IV heart failure, (2) unstable angina, (3) a history of recent (within 6 months) myocardial infarction or sustained (> 30 second) ventricular tachyarrhythmias, or (4) cerebrovascular accident
* Any active infection currently being treated or any infection within the last 6 weeks that required 7 days or more of IV antibiotics or any active infection within the last 4 weeks that requires use of oral antibiotics. Patients may be eligible once these timeframes elapse and with evidence that the infection has completely resolved
* Have inadequate venous access for or contraindications for the apheresis procedure
* Must agree not to participate in a conception process or must agree to a highly effective method of contraception

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
Dose Escalation: Dose Identification of CART-PSMA-TGFβRDN | Up to 2 years
  Incidence of Dose Limiting Toxicity (DLT)
Cohort Expansion: Safety of CART-PSMA-TGFβRDN | Up to 2 years
  Percentage of patients experiencing adverse events (AEs), including serious and severe AEs overall, by dose level, and severity grade

SECONDARY OUTCOMES:
Preliminary efficacy of CART-PSMA-TGFβRDN as assessed by biochemical Objective Response Rate (ORR) | Up to 2 years
  ORR defined as the proportion of patients with maximal prostate-specific antigen (PSA) decline of greater than or equal to 50% at 12 weeks post infusion
Feasibility of CART-PSMA-TGFβRDN | Up to 2 years
  Proportion of patients who did not receive CART-PSMA-TGFβRDN cells
Peripheral expansion and persistence of CART-PSMA-TGFβRDN | Up to 15 years
  Quantitative polymerase chain reaction (qPCR)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Moffitt Cancer Center, Tampa, Florida
  - The University of Kansas Hospital, Kansas City, Kansas
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Insitute, Nashville, Tennessee
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No